CLINICAL TRIAL: NCT04323956
Title: Phase I/Ib Study of Parsaclisib (INCB50465), Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone (PaR-CHOP) Immunochemotherapy for Patients With Newly Diagnosed High Risk Diffuse Large B-Cell Lymphoma
Brief Title: Parsaclisib Plus the Standard Drug Therapy in Patients With Newly Diagnosed, High Risk Diffuse Large B-cell Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC1986; NCI-2020-01855 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-005387 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Ann Arbor Stage II Diffuse Large B-Cell Lymphoma; Ann Arbor Stage II Follicular Lymphoma; Ann Arbor Stage II Marginal Zone Lymphoma; Ann Arbor Stage III Diffuse Large B-Cell Lymphoma; Ann Arbor Stage III Follicular Lymphoma; Ann Arbor Stage III Marginal Zone Lymphoma; Ann Arbor Stage IV Diffuse Large B-Cell Lymphoma; Ann Arbor Stage IV Follicular Lymphoma; Ann Arbor Stage IV Marginal Zone Lymphoma; Diffuse Large B-Cell Lymphoma; High Grade B-Cell Lymphoma With MYC and BCL2 and/or BCL6 Rearrangements; High Grade B-Cell Lymphoma With MYC and BCL2 or BCL6 Rearrangements; High Grade B-Cell Lymphoma With MYC, BCL2, and BCL6 Rearrangements; Indolent Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Cyclophosphamide; Doxorubicin; parsaclisib; pegfilgrastim; pegylated granulocyte colony-stimulating factor; polatuzumab vedotin; Prednisone; deltacortene; prednylidene; Rituximab; CT-P10; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (parsaclisib, R-CHOP) (Experimental): Patients receive parsaclisib PO QD on days 1-10 or 1-14, rituximab IV or biosimilar substitute, cyclophosphamide IV over 30 minutes, doxorubicin hydrochloride IV, and vincristine sulfate IV over 15 minutes on day 1. Patients also receive prednisone PO on days 1-5 and pegfilgrastim SC or biosimilar substitute on day 2. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Parsaclisib; Biological: Pegfilgrastim; Drug: Prednisone; Biological: Rituximab; Drug: Vincristine Sulfate
- Arm II (parsaclisib, R-CHOP, polatuzumab vedotin) (Active Comparator): Patients receive parsaclisib PO once daily QD on days 1-10 or 1-14, polatuzumab vedotin IV over 90 minutes, rituximab IV or biosimilar substitute, cyclophosphamide IV over 30 minutes, doxorubicin hydrochloride IV, and vincristine sulfate IV over 15 minutes on day 1. Patients also receive prednisone PO on days 1-5 and pegfilgrastim SC or biosimilar substitute on day 2. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Parsaclisib; Biological: Pegfilgrastim; Drug: Polatuzumab Vedotin; Drug: Prednisone; Biological: Rituximab; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719; Asta B 518; B-518; WR-138719
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Drug: Parsaclisib — Given PO
  Other Names: (4R)-4-(3-((1S)-1-(4-Amino-3-methyl-1H-pyrazolo(3,4-d)pyrimidin-1-yl)ethyl)-5-chloro-2-ethoxy-6-fluorophenyl)pyrrolidin-2-one; IBI376; INCB 50465; INCB-50465; INCB050465; INCB50465; WHO 10589
Biological: Pegfilgrastim — Given SC
  Other Names: Filgrastim SD-01; filgrastim-SD/01; Fulphila; HSP-130; Jinyouli; Neulasta; Neulastim; Nyvepria; PEG-filgrastim; Pegcyte; Pegfilgrastim Biosimilar HSP-130; Pegfilgrastim Biosimilar Nyvepria; Pegfilgrastim Biosimilar Pegcyte; Pegfilgrastim Biosimilar PF-06881894; Pegfilgrastim Biosimilar Udenyca; Pegfilgrastim Biosimilar Ziextenzo; pegfilgrastim-apgf; pegfilgrastim-bmez; pegfilgrastim-cbqv; Pegfilgrastim-jmdb; PF-06881894; SD-01; SD-01 sustained duration G-CSF; Udenyca; Ziextenzo; Neupopeg; Pegylated G-CSF; Pegylated GCSF; Pegylated Granulocyte Colony Stimulating Factor
Drug: Polatuzumab Vedotin — Given IV
  Other Names: ADC DCDS4501A; Antibody-Drug Conjugate DCDS4501A; DCDS4501A; FCU 2711; polatuzumab vedotin-piiq; Polivy; RG7596; Ro 5541077-000
  Arms: Arm II (parsaclisib, R-CHOP, polatuzumab vedotin)
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Riabni; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; rituximab-abbs; Rituximab-arrx; Rituximab-pvvr; RTXM83; Ruxience; Truxima; Ikgdar; Mabtas
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase I/Ib trial studies the side effects and best dose of parsaclisib with or without polatuzumab-vedotin (Pola) plus the standard drug therapy (rituximab, cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, and prednisone [PaR-CHOP]) and to see how well they work compared with R-CHOP alone in treating patients with newly diagnosed, high risk diffuse large B-cell lymphoma. Parsaclisib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Rituximab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Polatuzumab-vedotin is a monoclonal antibody, called polatuzumab, linked to a chemotherapy drug, called vedotin. Polatuzumab is a form of targeted therapy because it attaches to specific molecules (receptors) on the surface of cancer cells, known as anti-CD79b receptors, and delivers vedotin to kill them. Drugs used in chemotherapy, such as cyclophosphamide, doxorubicin hydrochloride, and vincristine sulfate, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Anti-inflammatory drugs, such as prednisone, lower the body's immune response and are used with other drugs in the treatment of some types of cancer. It is not yet known if giving parsaclisib and R-CHOP together works better than R-CHOP alone in treating patients with high risk diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the maximum tolerated dose (MTD) of parsaclisib in combination with R-CHOP in newly diagnosed diffuse large B-cell lymphoma (DLBCL). (Phase I) II. To assess the complete metabolic response rate by positron emission tomography (PET) (PET complete response [CR]) of combining parsaclisib and R-CHOP in patients with newly diagnosed DLBCL. (Dose Expansion) III. To assess significant toxicities of parsaclisib in combination with polatuzumab vedotin (pola) and R-CHP in newly diagnosed DLBCL. (Pola Safety Lead-in)

SECONDARY OBJECTIVES:

I. To describe the toxicities associated with parsaclisib in combination with R-CHOP. (Phase I) II. To assess the objective response rate (ORR) of parsaclisib in combination with R-CHOP. (Dose Expansion) III. To assess the duration of response (DOR), event-free survival (EFS), progression-free survival (PFS), and overall survival (OS) in patients treated with parsaclisib in combination with R-CHOP. (Dose Expansion) IV. To further describe the toxicities associated with parsaclisib in combination with R-CHOP. (Dose Expansion) V. To describe the toxicities associated with parsaclisib in combination with polatuzumab vedotin and R-CHP. (Pola Safety Lead-in) VI. To assess the PET CR rate and ORR of parsaclisib in combination with polatuzumab vedotin and R-CHP. (Pola Safety Lead-in) VII. To assess the duration of response (DOR), event-free survival (EFS), progression-free survival (PFS), and overall survival (OS) in patients treated with parsaclisib in combination with polatuzumab vedotin and R-CHP. (Pola Safety Lead-in)

OUTLINE: This is a phase I, dose-escalation study of parsaclisib, and safety lead-in of pola.

ARM I (PHASE I AND DOSE EXPANSION): Patients receive parsaclisib orally (PO) once daily (QD) on days 1-10 or 1-14, rituximab intravenously (IV) or biosimilar substitute, cyclophosphamide IV over 30 minutes, doxorubicin hydrochloride IV, and vincristine sulfate IV over 15 minutes on day 1. Patients also receive prednisone PO on days 1-5 and pegfilgrastim subcutaneously (SC) or biosimilar substitute on day 2. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

ARM II (PHASE I AND POLA SAFETY LEAD-IN): Patients receive parsaclisib PO once daily QD on days 1-10 or 1-14, polatuzumab vedotin IV over 90 minutes, rituximab IV or biosimilar substitute, cyclophosphamide IV over 30 minutes, doxorubicin hydrochloride IV, and vincristine sulfate IV over 15 minutes on day 1. Patients also receive prednisone PO on days 1-5 and pegfilgrastim SC or biosimilar substitute on day 2. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months during year 1 and every 4 months during year 2. Patients who experience disease progression before the end of year 2 are followed up every 6 months until 5 years after registration.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Newly diagnosed, untreated, histologically confirmed diffuse large B-cell lymphoma expressing the CD20 antigen, with ANY of the following:

  * Non-germinal center B-cell (GCB) subtype by Hans algorithm
  * Myc expression >= 40% by immunohistochemistry (IHC)
  * Bcl-2 expression >= 50% by IHC
  * Myc expression >= 40% AND Bcl-2 expression >= 50% by IHC (double expressor)
  * MYC rearrangement by fluorescence in situ hybridization (FISH)
  * Or high-grade B-cell lymphoma with MYC rearrangement AND BCL2 and/or BCL6 rearrangement (double-hit or triple-hit lymphoma) but not a candidate for more aggressive chemotherapy (such as cyclophosphamide, Oncovin [vincristine], doxorubicin, [CODOX]-methotrexate [M]- ifosfamide, Vepesid [etoposide], Ara-C [cytarabine] [IVAC])

    * NOTE: Patients with a new diagnosis of concurrent DLBCL and an indolent lymphoma (previously undiagnosed, such as follicular lymphoma or marginal zone lymphoma) are eligible. However, patients with a known prior diagnosis of indolent lymphoma with new transformation to DLBCL (i.e., transformed lymphoma) are not eligible
* Ann Arbor stages II (bulky disease, i.e., >= 5 cm, or not a candidate for combined modality treatment with R-CHOP plus radiotherapy), III, or IV
* Measurable disease (at least 1 lesion of >= 1.5 cm in one diameter) as detected by computed tomography (CT) or the CT images of PET/CT. Skins lesions can be used if the area is >= 2 cm in at least one diameter and photographed with a ruler
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Absolute neutrophil count (ANC) >= 1500/mm^3 (obtained =< 14 days prior to registration)
* Platelet count >= 100,000/mm^3 (obtained =< 14 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN), or if total bilirubin is > 1.5 x ULN, the direct bilirubin must be normal (obtained =< 14 days prior to registration)
* Aspartate transaminase (AST) =< 3 x ULN (=< 5 x ULN for patients with direct liver involvement by lymphoma) (obtained =< 14 days prior to registration)
* Alkaline phosphatase =< 3 x ULN, unless evidence of the direct liver involvement by lymphoma, then =< 5 x ULN (obtained =< 14 days prior to registration)
* Calculated creatinine clearance of >= 30 mL/min using the Cockcroft-Gault formula (obtained =< 14 days prior to registration)
* Negative urine pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only

  * NOTE: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Persons of childbearing potential must agree to use one reliable form of birth control
* Provide written informed consent
* Willingness to provide mandatory research blood specimens for banking
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)

Exclusion Criteria:

* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant persons
  * Nursing persons (lactating persons are eligible provided that they agree not to breast feed while taking parsaclisib)
  * Persons of childbearing potential who are unwilling to employ adequate contraception
* Primary central nervous system (CNS) lymphoma, or parenchymal, meningeal or cerebrospinal fluid involvement with malignant lymphoma cells
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy (except for patients on effective antiretroviral therapy with undetectable viral load within 6 months)

  * NOTE: If evidence of chronic hepatitis B virus (HBV) infection, HBV viral load must be undetectable on suppressive therapy if indicated
  * NOTE: If history of hepatitis C virus (HCV) infection, HCV viral load must be undetectable
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Ongoing inflammatory bowel disease (such as ulcerative colitis) or other colitis requiring active treatment
  * Oxygen dependent baseline lung disease (such as interstitial lung disease or chronic obstructive pulmonary disease [COPD])
  * Or psychiatric illness/social situations that would limit compliance with study requirements
* Received or receiving any other agent which would be considered as a treatment for the lymphoma (with the exception of corticosteroid)
* Other active malignancy requiring therapy such as radiation, chemotherapy or immunotherapy. Patients on hormonal therapy for treated breast or prostate cancer are permitted if they meet other eligibility criteria

  * EXCEPTIONS: Localized non-melanotic skin cancer or any cancer that in the judgment of the investigator has been treated with curative intent (e.g., disease-free survival equal or more than 5 years) and will not interfere with the study treatment plan and response assessment
  * NOTE: If there is a history of prior malignancy, they must not require therapy such as radiation, chemotherapy or immunotherapy for their cancer
* History of myocardial infarction =< 6 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* >= 25% of bone marrow radiated for other diseases
* Ejection fraction of < 45% by either multigated acquisition scan (MUGA) or echocardiogram (ECHO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2028-05-16 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of parsaclisib in combination with rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP) (Phase I) | Up to 21 days
  The MTD will be defined as the dose level below the lowest dose that induces dose-limiting toxicity in in at least one-third of patients (at least 2 of a maximum of 6 patients).
Complete metabolic response (CMR) rate (Dose Expansion) | Up to end of treatment (3-4 weeks after day 1 of cycle 6 [each cycle is 21 days])
  Will be measured by positron emission tomography (PET). A success is defined as an objective status of CMR by the PET-computed tomography (CT) based response criteria at the end of treatment. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true rate of complete metabolic response will be calculated.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) (Phase I) | Up to 2 years
  The number and severity (grade) of all treatment related AEs will be tabulated and summarized. Non-hematologic AEs will be evaluated via the ordinal Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0 standard AE grading. Hematologic toxicity measures of thrombocytopenia, neutropenia, and leukopenia will be assessed using continuous variables as the outcome measures (primarily nadir) as well as categorization via CTCAE v 5.0 standard AE grading. Both all grade and grade 3 and above AEs will be described and summarized in a similar fashion. Overall AE incidences as well as AE profiles by dose level and patient will be explored and summarized. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses.
Incidence of toxicity due to parsaclisib in combination with Pola-R-CHP (Pola Safety Lead-in) | Up to cycle 1 (21 days)
  Toxicity will be measured per NCI-CTCAE version 5. Significant toxicity is defined as an adverse event occurring during the first cycle of treatment that is possibly, probably, or definitely related to study treatment.
Objective response rate (Dose Expansion) | Up to end of treatment (3-4 weeks after day 1 of cycle 6 [each cycle is 21 days])
  Will be estimated by the number of patients with an objective status of CMR or partial metabolic response (PMR) by the PET-CT based response criteria at the end of treatment divided by the total number of evaluable patients. All evaluable patients will be used for this analysis. Exact binomial 95% confidence intervals for the true objective response rate will be calculated.
Duration of response (Dose Expansion) | Up to 2 years
  Defined as the date at which the patient's objective status is first noted to be either CMR or PMR to the earliest date progression is documented by CT or PET/CT [progressive metabolic disease (PMD) or progressive disease (PD)]
Event-free survival (Dose Expansion) | Up to 5 years
  Defined as the time from registration to disease progression or relapse (PMD or PD), initiation of subsequent anti-lymphoma therapy, or death due to any cause.
Progression-free survival (Dose Expansion) | Up to 5 years
  Defined as the time from registration to progression (PMD or PD) or death due to any cause
Overall survival (Pola Safety Lead-in) | Up to 5 years
  Defined as the time from registration until death due to any cause.
Incidence of adverse events (Dose Expansion) | Up to 2 years
  The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration.
Objective response rate (Pola Safety Lead-in) | Up to end of treatment [3-4 weeks after day 1 of cycle 6 (each cycle is 21 days)]
  Will be estimated by the number of patients with an objective status of CMR or PMR by the PET-CT based response criteria at the end of treatment divided by the total number of evaluable patients. All evaluable patients will be used for this analysis. Exact binomial 95% confidence intervals for the true objective response rate will be calculated.
Duration of response (Pola Safety Lead-in) | Up to 2 years
  Defined as the date at which the patient's objective status is first noted to be either CMR or PMR to the earliest date progression is documented by CT or PET/CT (PMD or PD)
Event-free survival (Pola Safety Lead-in) | Up to 5 years
  Defined as the time from registration to disease progression or relapse (PMD or PD), initiation of subsequent anti-lymphoma therapy, or death due to any cause
Progression-free survival (Pola Safety Lead-in) | Up to 5 years
  Defined as the time from registration to progression (PMD or PD) or death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Yucai Wang, M.D., Ph.D., Principal Investigator — Mayo Clinic in Rochester
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials